CLINICAL TRIAL: NCT03583138
Title: Project STRIDE2 - Seek/Test/Retain: PLWHA and Opioid Users in Washington, DC
Brief Title: HIV, Buprenorphine, and the Criminal Justice System (STRIDE2)
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); George Mason University (Other); Howard University (Other)
Responsible Party: Sponsor
Other Study IDs: 1011007631b; R01DA030768 (NIH)
Record Dates: First submitted 2018-03-19; First posted 2018-07-11 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Human Immunodeficiency Virus; Acquired Immunodeficiency Syndrome; Opiate Addiction; Drug Dependence
Keywords: HIV; AIDS; Opiate Addiction; Drug Dependence; Buprenorphine
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Opioid-Related Disorders; Substance-Related Disorders | interventions — Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Buprenorphine: Participants are eligible for the study if they are 18 years of age or older, HIV+, meet DSM-IV criteria for opioid dependence, have health insurance accepted at Lab Corp, are able to read and understand English, and live in Washington, DC and plan to remain in DC. The intervention is to provide buprenorphine for 12 months for those who are interested in receiving it.
  Interventions: Drug: buprenorphine
- No buprenorphine: No buprenorphine

INTERVENTIONS:
Drug: buprenorphine — To provide buprenorphine for 12 months for those who are interested in receiving it.
  Other Names: Suboxone
  Groups: Buprenorphine

SUMMARY:
STRIDE2 is a longitudinal, non-randomized study of individuals living with HIV who are dependent on opioids. This study is funded by the National Institute on Drug Abuse (R01DA030768, Altice, PI; Taxman & Lawson, Co-PIs) and is being conducted by George Mason University, Yale University, and Howard University.

DETAILED DESCRIPTION:
STRIDE2 will assist in identifying and monitoring individuals' HIV risk behaviors and provide resources to seek treatment for their HIV care and substance use. The goal of STRIDE2 is to examine if there are differences in HIV, drug use, and other outcomes between individuals receiving treatment versus individuals actively using, not actively using and not in treatment, and individuals on Methadone, Suboxone, or in some other treatment.

ELIGIBILITY:
Inclusion Criteria:

1. HIV+, confirmed by rapid HIV test
2. Meet DSM-IV criteria for opioid dependence
3. 18 years or older
4. Have health insurance that is accepted at Lab Corp.

Exclusion Criteria:

1. Are <18 years old;
2. Are HIV negative;
3. Are Unable to communicate in English;
4. Are not able to provide informed consent;
5. Do not meet DSM-IV criteria for opioid dependence;
6. Plan to leave the DC area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years of age or older, HIV+, meet DSM-IV criteria for opioid dependence, have health insurance accepted at Lab Corp, are able to read and understand English, and live in Washington, DC and plan to remain in DC.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2014-06-23 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
VL <400 | Month 0
  Blood test for HIV viral load
CD4+ cell count | Month 0
  Blood test for HIV CD4+ cell count
VL <400 | 6 months
  Blood test for HIV viral load
CD4+ cell count | 6 months
  Blood test for HIV CD4+ cell count
VL <400 | 12 months
  Blood test for HIV viral load
CD4+ cell count | 12 months
  Blood test for HIV CD4+ cell count

SECONDARY OUTCOMES:
HIV risk behaviors | Month 0
  Survey for HIV risks
HIV risk behaviors | 6 months
  Survey for HIV risks
HIV risk behaviors | 12 months
  Survey for HIV risks
Retention in HIV care | Month 0
  Survey data for retention
Retention in HIV care | 6 months
  Survey data for retention
Retention in HIV care | 12 months
  Survey data for retention
Opioid use | Month 0
  Measure of relapse to opioid use
Opioid use | 6 months
  Measure of relapse to opioid use
Opioid use | 12 months
  Measure of relapse to opioid use
Medically assisted therapy retention | Month 0
  Measure of length of time on Methadone or Buprenorphine
Medically assisted therapy retention | 6 months
  Measure of length of time on Methadone or Buprenorphine
Medically assisted therapy retention | 12 months
  Measure of length of time on Methadone or Buprenorphine

OTHER OUTCOMES:
Reincarceration | Month 0
  Measure of rearrest and reincarceration
Reincarceration | 6 months
  Measure of rearrest and reincarceration
Reincarceration | 12 months
  Measure of rearrest and reincarceration

CONTACTS AND LOCATIONS:
Overall Officials: Fredrick Altice, MD, Principal Investigator — Yale University School of Medicine/AIDS Program; Faye Taxman, PhD, Principal Investigator — George Mason University; William Lawson, MD, Principal Investigator — Howard University
Locations (1):
- Howard University, Washington D.C., District of Columbia, United States